CLINICAL TRIAL: NCT06796465
Title: Effects of Mckenzie Protocol With and Without Progressive Postural Control Exercise on Pain, Range of Motion and Disability in Patients With Low Back Pain
Brief Title: McKenzie Protocol With/Without Postural Control Exercises on Pain, ROM, and Disability in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0122
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain
Keywords: Low back pain; McKenzie exercise; Progressive postural control exercise
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A received a combination of McKenzie exercises and Progressive Postural Control Exercises. Each session began with the application of hot packs for 10-15 minutes to prepare the patients for the exercises. Patients then performed three sets of three exercises, with 10 repetitions per set, lasting approximately 10-15 minutes in total.
  Interventions: Other: McKenzie with Progressive Postural Control Exercises; Device: Hot Pack
- Group B (Experimental): Group B was treated with McKenzie exercises without the integration of Progressive Postural Control Exercises. Each session began with the application of hot packs for 10-15 minutes to prepare the patients for the technique. Patients then performed three sets of three exercises, with 10 repetitions per set, lasting approximately 10-15 minutes in total.
  Interventions: Other: McKenzie without Progressive Postural Control Exercises; Device: Hot Pack

INTERVENTIONS:
Other: McKenzie with Progressive Postural Control Exercises — The McKenzie Exercises focus on progressive spinal extension to alleviate back pain. Key steps include Extension in Standing, where patients lean backward and return to a neutral stance; Extension in Lying (Partial Range), involving partial pushups in a prone position; and Extension in Lying (Full Range), where patients fully extend their arms to achieve maximum spinal extension. Each movement is held for 1-2 seconds.
  The PPCE program enhances core strength and stability through three stages. In the First Stage (2 weeks), core muscles are trained against gravity using movements like pelvic retroversion, crunches, and glute bridges. The Second Stage (3 weeks) incorporates a Swiss ball to challenge trunk muscles with instability. In the Third Stage (3 weeks), a Swiss ball, stretch bands, and a 5 kg sandbag are used to increase complexity on unstable surfaces. Each stage includes six movements, lasting 5 minutes each, for a total session duration of 30 minutes.
  Other Names: McKenzie; Progressive Postural Control
  Arms: Group A
Other: McKenzie without Progressive Postural Control Exercises — Subject were treated with McKenzie exercises without the addition of Progressive Postural Control Exercises (PPCE).The exercises included the following:
  Standing Extension Exercises: Patients leaned backward from a balanced standing position, arching their back before returning to a neutral stance.
  Extension in Lying (Partial Range): Performed in a prone position with hands placed under the shoulders, patients lifted their upper torso in a motion similar to a push-up.
  Extension in Lying (Full Range): Similar to the partial range extension, but with fully extended arms, aiming for the maximum tolerated extension. Each movement was sustained for 1-2 seconds.
  Arms: Group B
Device: Hot Pack — for 10 to 15 minutes

SUMMARY:
Chronic Low Back Pain (CLBP) is a prevalent global musculoskeletal disorder associated with significant physical, psychosocial, and economic burdens. The McKenzie method focuses on the use of sustained postures or repeated movements tailored to alleviate pain and restore function. Progressive Postural Control Exercise (PPCE) is an innovative approach for managing CLBP. It combines elements of motor control exercises and resistance training, emphasizing challenges to postural control through phased progression to improve stability and function.

The aim of this study is to compare the effects of the McKenzie protocol, both with and without the integration of Progressive Postural Control Exercises (PPCE), on pain, range of motion, and disability in patients with low back pain.

This study utilized a randomized controlled design with two groups. Participants were recruited from Shaikh Zaid Hospital using non-probability convenience sampling. The intervention lasted six weeks, with assessments conducted at baseline, three weeks, and six weeks.

Group A received McKenzie exercises combined with Progressive Postural Control Exercises (PPCE), while Group B was treated with McKenzie exercises alone, without PPCE. Assessment tools included the Numeric Pain Rating Scale (NPRS) for pain, the Roland-Morris Disability Questionnaire (RMDQ) for disability, the Oswestry Disability Index (ODI) for disability, and an inclinometer for measuring range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* Diagnosed with non-specific low back pain, with symptoms and pain persisting for over 3 months
* Individuals reporting a pain intensity of at least 4 out of 7 on the 11-point Numeric Pain Rating Scale (11-NPRS)
* Individuals scoring 4 or above on the Roland-Morris Questionnaire (RMQ) for low back pain

Exclusion Criteria:

* Pregnancy
* Chronic low back pain (LBP) due to trauma, structural issues, neurological symptoms, or radiating pain to the lower legs
* History of back surgery, spinal tumors, or infections
* Diagnosed neurological or musculoskeletal disorders unrelated to LBP, including, Stroke, Parkinson's disease, Demyelination disorders, Multiple sclerosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-02-11 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
NPRS | Baseline, 3 and 6 weeks
  The Numeric Pain Rating Scale (NPRS) will be used to assess patients' pain levels for chronic low back pain both before and after the exercises. This 11-point numeric scale ranges from 0, representing no pain (e.g., "no pain at all"), to 10, representing the worst pain imaginable (e.g., "pain as bad as you can imagine" or "worst pain imaginable"). The NPRS demonstrates strong validity, with values ranging from 0.86 to 0.96
The Roland-Morris Disability Questionnaire | Baseline, 3 and 6 weeks
  The Roland-Morris Disability Questionnaire (RMDQ) is a reliable and widely used tool for assessing disability in patients with low back pain. Its updated applications and adaptations have reinforced its validity across diverse patient populations and healthcare settings. The RMDQ consists of 24 items, with the total score calculated by summing the responses. A "yes" response is scored as 1, and a "no" response is scored as 0, resulting in a total score range of 0 to 24. This range reflects the level of disability, with higher scores indicating greater disability in individuals with low back pain.

SECONDARY OUTCOMES:
Inclinometer | Baseline, 3 and 6 weeks
  The inclinometer is a widely used tool in clinical and research settings for measuring the range of motion (ROM) in spinal, cervical, and limb assessments. It is particularly valuable in managing conditions such as thoracic kyphosis and general musculoskeletal dysfunction. The device demonstrates excellent reliability, with inter-rater correlation coefficients (ICC) around 0.96, indicating high agreement and consistency between different raters.

CONTACTS AND LOCATIONS:
Overall Officials: Humera Mubashar, MS OMPT, Principal Investigator — Riphah International University
Locations (1):
- Shaikh Zayed Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang H, Fan Z, Liu X, Zheng J, Zhang S, Zhang S, Yu Q, Lo WLA, Chen X, Wang C. Effect of Progressive Postural Control Exercise Versus Core Stability Exercise in Young Adults with Chronic Low Back Pain: A Randomized Controlled Trial. Pain Ther. 2023 Feb;12(1):293-308. doi: 10.1007/s40122-022-00458-x. Epub 2022 Dec 1. PMID 36454387